CLINICAL TRIAL: NCT07248020
Title: A Phase II Single-Arm Study of High-Bioavailability Curcumin as Neoadjuvant Chemoradiotherapy in Mid-to-Low Rectal Cancer: Integrated Clinical and Translational Analysis of Tumor Tissue
Acronym: BCMRECRAD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202501055A0
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Rectal Cancer; Locally Advanced Rectal Cancer; Radiation-Induced Enteritis; Radiation Proctitis; Chemoradiotherapy-Related Toxicity
Keywords: Curcumin; Rectal cancer; Chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label, phase II interventional study designed to evaluate the safety, tolerability, and therapeutic potential of high-bioavailability curcumin (BCM-95®) administered concurrently with standard neoadjuvant chemoradiotherapy (nCRT) in patients with mid-to-low rectal adenocarcinoma. All participants will receive oral BCM-95® (3 g/day) throughout the entire nCRT period.
  The study begins with a safety run-in cohort of six patients to confirm dose feasibility and monitor dose-limiting toxicities (DLTs), followed by expansion to a total of 72 patients. The intervention model follows a single-group assignment without randomization or masking. Outcomes include radiation-induced gastrointestinal toxicity, treatment completion, and tumor response. Translational analyses on serial tumor and blood samples will explore curcumin's anti-inflammatory and anti-cancer mechanisms.
Masking Description: This study is conducted as an open-label, single-arm trial. Because the investigational product (oral high-bioavailability curcumin, BCM-95®) is administered as a dietary supplement in combination with standard neoadjuvant chemoradiotherapy, blinding of participants and investigators is not feasible. The intervention does not involve a placebo or comparator arm, and all participants receive the same standardized treatment regimen. Safety, efficacy, and translational endpoints will be objectively assessed using predefined clinical and laboratory criteria (CTCAE v5.0, RTOG/EORTC, RECIST v1.1).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-Bioavailability Curcumin (BCM-95®) Plus Neoadjuvant Chemoradiotherapy (Experimental): Participants with stage II-III mid-to-low rectal adenocarcinoma will receive oral high-bioavailability curcumin (BCM-95®) 3 g per day throughout the entire course of standard neoadjuvant chemoradiotherapy (nCRT).
  nCRT will include:
  Short-course radiotherapy: 25 Gy in 5 fractions with systemic chemotherapy as per institutional protocol.
  Curcumin administration starts on the first day of chemoradiotherapy and continues until completion. The aim is to evaluate whether curcumin reduces radiation-induced gastrointestinal toxicity (enteritis/proctitis), enhances tumor response, and improves treatment tolerability. Translational analyses of tumor and blood samples will explore curcumin's anti-inflammatory and anti-cancer molecular mechanisms.
  Interventions: Dietary Supplement: Curcumin (BCM-95®)

INTERVENTIONS:
Dietary Supplement: Curcumin (BCM-95®) — Participants will receive oral high-bioavailability curcumin (BCM-95®) 3 g per day, divided into two doses, during the full course of standard neoadjuvant chemoradiotherapy (nCRT) for mid-to-low rectal adenocarcinoma. Treatment starts on day one of nCRT and continues until its completion.
  The curcumin formulation (BCM-95®) combines curcuminoids with turmeric essential oils to improve systemic absorption and bioavailability. All participants receive institutional standard nCRT, including:
  Radiotherapy: either long-course (50.4 Gy/28 fractions) or short-course (25 Gy/5 fractions).
  Chemotherapy: fluoropyrimidine-based regimens such as TEGAFOX, FOLFOX, or UFUR.
  Curcumin capsules are taken orally after meals. The study evaluates whether curcumin can reduce radiation-induced gastrointestinal toxicity and enhance tumor response. Translational analyses of tumor and blood samples will further investigate its anti-inflammatory and anti-cancer mechanisms.
  Other Names: High-Bioavailability Curcumin; BCM95 Curcumin

SUMMARY:
This clinical study investigates the anti-inflammatory and anti-cancer properties of a high-bioavailability formulation of curcumin (BCM-95) in patients with mid-to-low rectal cancer receiving neoadjuvant chemoradiotherapy (nCRT). Curcumin, a polyphenolic compound derived from Curcuma longa, has demonstrated potent anti-inflammatory and anti-neoplastic activities through the modulation of multiple molecular signaling pathways. It has been recognized by the U.S. Food and Drug Administration (FDA) as "Generally Recognized as Safe" (GRAS; GRN No. 686), with an excellent safety profile when administered orally. Reported adverse effects are rare and primarily related to interference with bile secretion or iron metabolism.

Despite its biological potential, conventional curcumin exhibits extremely low oral bioavailability due to its lipophilic nature, rapid metabolism, and systemic elimination. Clinical studies have reported that even at an oral dose of 12 grams per day, the maximum plasma concentration reaches only about 0.051 mg/mL, with up to 75% of the administered dose excreted in feces. To overcome this limitation, the current trial utilizes a curcumin formulation with enhanced absorption (BCM-95), which combines curcumin with essential oils of turmeric to improve systemic bioavailability.

The primary objective of this single-arm, phase II trial is to evaluate whether oral curcumin supplementation can mitigate radiation-induced gastrointestinal toxicity-particularly radiation enteritis-during neoadjuvant chemoradiotherapy for rectal cancer. The secondary objectives include assessing its effect on treatment response, such as the pathological complete response (pCR) rate, tumor regression grade, and patient-reported outcomes related to bowel function and quality of life.

In addition, a translational research component is embedded within this study. Serial tumor tissue and blood samples will be collected at predefined time points to explore the molecular and immunological mechanisms underlying curcumin's therapeutic effects. Analyses will include assessments of inflammatory cytokines, oxidative stress markers, and tumor microenvironmental changes using molecular and histopathologic methods.

Overall, this study aims to provide both clinical and mechanistic evidence supporting the potential of high-bioavailability curcumin as a safe, adjunctive therapeutic strategy to improve treatment tolerance and oncologic outcomes in rectal cancer patients undergoing chemoradiotherapy.

DETAILED DESCRIPTION:
This Phase II single-arm clinical trial investigates the safety, tolerability, and therapeutic potential of high-bioavailability curcumin (BCM-95®) administered concurrently with neoadjuvant chemoradiotherapy (nCRT) in patients with mid- to low-rectal adenocarcinoma. The study is designed and conducted at Chang Gung Memorial Hospital, Linkou (Taiwan), under IRB approval and in accordance with Good Clinical Practice (GCP) guidelines.

Scientific Background and Rationale

Curcumin (diferuloylmethane) is a hydrophobic polyphenol extracted from Curcuma longa with extensive anti-inflammatory, antioxidant, and anti-neoplastic properties mediated through suppression of NF-κB, STAT3, COX-2, and multiple cell-signaling pathways. In preclinical models, curcumin inhibits radiation-induced activation of NF-κB and enhances radiosensitivity of colorectal-cancer cell lines, while protecting normal intestinal epithelium from irinotecan-induced mucosal injury by mitigating oxidative and endoplasmic-reticulum stress. Despite its excellent oral safety record (FDA GRAS Notice No. 686), conventional curcumin suffers from extremely low systemic bioavailability due to poor solubility and rapid metabolism.

BCM-95® Curcumin is a patented formulation that combines 95 % curcuminoids with turmeric essential oils, improving absorption approximately seven-fold compared with standard curcumin. Given its dual ability to radiosensitize tumor tissue and protect normal mucosa, BCM-95® Curcumin may attenuate radiation-induced enteritis while enhancing tumor regression and pathological complete-response (pCR) rates following nCRT.

Objectives

Primary Objective: To evaluate whether oral BCM-95® Curcumin can reduce the incidence and severity of radiation-induced gastrointestinal toxicity, particularly grade ≥ 3 proctitis/enteritis, during nCRT.

Secondary Objectives: To assess improvement in treatment response (clinical and pathological CR rates, tumor-regression grade), treatment completion rate, and quality-of-life indices; and to explore anti-cancer and immunomodulatory mechanisms through translational analyses of tumor and blood specimens.

Study Overview

A total of 72 patients with stage II-III (mid- to low-) rectal adenocarcinoma will receive standard long-course nCRT (50.4 Gy in 28 fractions with concurrent fluoropyrimidine-based chemotherapy) or equivalent short-course radiotherapy plus chemotherapy, along with oral BCM-95® Curcumin 3 g per day. Treatment begins concurrently with chemotherapy and continues through the full nCRT period. Follow-up includes surgical resection or a watch-and-wait strategy based on clinical response.

Each participant undergoes serial evaluations:

Baseline: history, colonoscopy, pelvic MRI, CT staging, laboratory profile, and CEA.

During therapy: bi-weekly hematology and biochemistry tests; adverse-event assessment (CTCAE v5.0, RTOG/EORTC criteria).

Post-radiation (2-3 weeks): colonoscopy graded by Vienna Rectoscopy Score to quantify acute proctitis.

At completion of nCRT: pelvic MRI and colonoscopy for clinical response evaluation.

Surgery or watch-and-wait: histopathologic examination for pCR and tumor-regression grade.

Translational research includes multiplex immunohistochemistry on paired tumor and adjacent mucosa (pre-treatment, post-radiation, post-CRT) and peripheral-blood analyses for immune-cell phenotyping (BD FACSymphony panel), cytokine profiling (MILLIPLEX array), and circulating-tumor-DNA (ctDNA) monitoring. These studies aim to correlate molecular and immune alterations with clinical outcomes.

Run-in Cohort (Safety Lead-in)

A run-in phase enrolling 6 patients will precede full recruitment. Dose-limiting toxicities (DLTs) include grade ≥ 3 non-hematologic AEs (except expected nausea/vomiting), ALT/AST > 3×ULN (confirmed) or > 5×ULN any time, bilirubin > 2×ULN with hepatic enzyme elevation, grade 4 hematologic toxicity > 7 days, or any toxicity requiring treatment interruption > 2 weeks. If ≤ 1/6 patients develops a DLT, the study proceeds to full Phase II enrollment (n = 72).

Endpoints

Primary Endpoint: Incidence of grade ≥ 3 gastrointestinal toxicity (enteritis/proctitis) evaluated by NCI CTCAE v5.0 and RTOG/EORTC criteria.

Secondary Endpoints: (1) Vienna Rectoscopy Score; (2) any grade III AEs during therapy; (3) clinical CR rate (RECIST v1.1); (4) pathological CR rate; (5) treatment completion rate.

Exploratory Endpoints: three-year disease-related failure rate, five-year overall survival, and molecular/immunologic correlates.

Statistical Considerations

The sample size (n = 72, 64 evaluable) was calculated by an exact one-proportion test (80 % power, α = 0.05) to detect a 15 % absolute reduction in acute radiation proctitis (30 % → 15 %). Efficacy and safety analyses follow the intent-to-treat principle. Categorical variables will be analyzed by χ² or Fisher's exact test; continuous variables by t or Mann-Whitney U test; survival by Kaplan-Meier and log-rank tests (p < 0.05 two-sided). Analyses will be performed in SPSS v24.

Safety Monitoring and Ethics

Safety is assessed continuously through bi-weekly labs and AE documentation. Curcumin is paused if ALT/AST > 3×ULN until recovery. Serious adverse events (SAEs) are reported to the Chang Gung IRB per institutional policy. The study follows the Declaration of Helsinki and GCP standards. All participants provide written informed consent. Confidentiality is maintained via coded identifiers; data access is restricted to authorized investigators.

Data and Safety Monitoring Plan (DSMP)

Enrollment review every 3 months by PI.

SAE review quarterly by Safety Officer.

Protocol deviation audit monthly by Clinical Research Coordinator.

Data integrity checked continuously by Data Manager. All findings are reported to the sponsor and IRB.

Anticipated Impact

This study will provide clinical and molecular evidence for the potential of high-bioavailability curcumin as a safe adjunct to neoadjuvant chemoradiotherapy in rectal cancer, with the dual goals of reducing treatment-related toxicity and enhancing tumor response and long-term oncologic outcomes. If proven beneficial, curcumin could be a cost-effective, natural, and readily implementable adjuvant strategy for improving tolerance and quality of life in rectal cancer patients undergoing multimodality therapy.

ELIGIBILITY:
Inclusion Criteria:

(A) Males and females more than 20 years of age (B) Signed informed consent (C) Patients with a pathologically proven rectal adenocarcinoma located less than 10 cm to the anus.

(D) Clinical staging (AJCC 8th ed.): T2-4 N0 M0 or T any N1-2 M0 (E) Distal metastasis has been excluded by imaging study: by chest-to-pelvic computed tomography or Positron Emission Tomography (F) Preoperative pelvic staging by pelvic Magnetic Resonance Imaging (preferred) or trans-rectal ultrasound (G) Patients with WHO/ECOG performance scale 0 or 1

Exclusion Criteria:

(A) Refuse to sign the informed consent (B) Distal metastasis revealed by the imaging study (C) Patients does not receive radiotherapy (D) Unable to receive further curative resection (E) Patients receive tumor resection before the neoadjuvant treatment (F) Patients have history of more than 5 Gy of pelvic radiation (G) Patients in pregnancy or lactation status (H) Patients have allergic history to curcumin, 5-fluouracil or oxaliplatin (I) Patients of childbearing potential can not cooperate with appropriate contraceptive method (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) (J) Patients with any concurrent malignancy; patients with history of malignancy should be cancer-free for more than 5 years (K) Patients with New York Heart Association (NYHA) class III or IV heart failure, unstable angina pectoris, unstable cardiac arrhythmia or tachycardia (heart rate > 100 beats/minute) (L) Patients have concurrent uncontrolled medical conditions, such as illness ongoing or requiring IV antibiotics, severe chronic renal failure (eGFR <30 mL/min/1.73m2) or severe active hepatitis(AST/ALT>3x upper normal limit)、Total Bilirubin>2 mg/dl (M) Patients with previous or current drug abuse (N) Patients underwent major surgery within 28 days of study enrollment (except diverting colostomy) (O) Patients have Familial Adenomatosis Polyposis Coli (FAP), Hereditary Non-Polyposis Colorectal Cancer (HNPCC), active Crohn's disease or active ulcerative Colitis (P) Patients have known dipyrimidine dehydrogenase deficiency (DPD) (Q) Patients with congenital iron metabolic or hematopoietic diseases (R) Patients with synchronous colon cancer (S) The Patients with hematologic abnormalities (INR > 1.5, white blood cell (WBC) count < 3,000/μL, absolute neutrophil count (ANC) < 1,500/μL, platelet count < 100,000/μL, hemoglobin < 9.0 g/dL not caused by tumor treatment) or known hematologic diseases (aplastic anemia, myelodysplastic syndrome (MDS), leukemia, malignant lymphoma, multiple myeloma, hereditary hematologic diseases such as thalassemia, sickle cell anemia, etc.).

(T) The patient has diabetes mellitus (U) The patient is taking the immunosuppressants Cyclosporine, Tacrolimus, Sirolimus, and Everolimus and antigoagulants (warfarin、NOACs、aspirin) (V) Patients with The medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade ≥3 Gastrointestinal Toxicity (Enteritis or Proctitis) During Neoadjuvant Chemoradiotherapy | From the start of chemoradiotherapy to 3 weeks after completion of radiotherapy (approximately 8 weeks total)
  The primary endpoint is the incidence of grade ≥3 gastrointestinal adverse events, including enteritis or proctitis, occurring during neoadjuvant chemoradiotherapy (nCRT). Toxicities will be assessed and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, and validated by Radiation Therapy Oncology Group (RTOG) and European Organisation for Research and Treatment of Cancer (EORTC) criteria. Clinical symptoms (abdominal pain, diarrhea, bloody stool, tenesmus, nausea) will be documented by investigators and research nurses. Colonoscopic assessment using the Vienna Rectoscopy Score will be performed 2-3 weeks after radiotherapy completion to evaluate acute radiation proctitis.

SECONDARY OUTCOMES:
Vienna Rectoscopy Score for Radiation-Induced Proctitis | Baseline, 2 ± 1 weeks, and 12 ± 1 weeks after completion of radiotherapy
  Endoscopic evaluation of rectal mucosa using the Vienna Rectoscopy Score (VRS) to assess the severity of radiation-induced proctitis. Colonoscopy will be performed before treatment, and again 2 ± 1 weeks and 12 ± 1 weeks after completion of radiotherapy. Scores will be compared across time points to determine curcumin's protective effect against radiation injury.

OTHER OUTCOMES:
Three-Year Disease-Related Treatment Failure Rate | From completion of chemoradiotherapy to 3 years after surgery
  Disease-related treatment failure is defined as the occurrence of any locoregional recurrence, distant metastasis, or cancer-related death from the completion of neoadjuvant chemoradiotherapy to three years after curative surgery. Disease status will be assessed through regular clinical visits, imaging studies (CT or MRI), and colonoscopic surveillance.
Five-Year Overall Survival | From the start of chemoradiotherapy to 5 years post-treatment
  Overall survival (OS) is defined as the time from the initiation of chemoradiotherapy to death from any cause. Patients will be followed through outpatient visits, hospital records, and national death registry data to determine long-term survival outcomes associated with curcumin treatment.
Molecular and Immune Marker Changes in Tumor and Adjacent Tissues | Baseline, post-radiotherapy (approximately 6 weeks), and at surgery (approximately 16-20 weeks after treatment start)
  Tumor and adjacent mucosal biopsies collected at baseline, after radiotherapy, and at surgery will be analyzed by multiplex immunohistochemistry to assess immune-cell infiltration (CD4⁺, CD8⁺ T cells, macrophages, dendritic cells) and expression of immune checkpoint molecules (PD-1, PD-L1, CTLA-4, CD47). Comparisons will determine how curcumin modulates the tumor microenvironment and inflammatory response.
Cytokine Profile and Circulating Tumor DNA (ctDNA) Dynamics | Baseline, after completion of chemoradiotherapy, and at surgery
  Peripheral blood samples will be analyzed for serum cytokines (Milliplex Human Cytokine/Chemokine Magnetic Bead Panel) and circulating tumor DNA (ctDNA) levels before and after neoadjuvant treatment. Changes in inflammatory cytokines and ctDNA concentration will be correlated with clinical and pathological response to curcumin-based therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Huan Huang, MD., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan District, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be shared because of patient privacy and institutional policy.

REFERENCES:
- [Result] Ouyang M, Luo Z, Zhang W, Zhu D, Lu Y, Wu J, Yao X. Protective effect of curcumin against irinotecan-induced intestinal mucosal injury via attenuation of NF-kappaB activation, oxidative stress and endoplasmic reticulum stress. Int J Oncol. 2019 Apr;54(4):1376-1386. doi: 10.3892/ijo.2019.4714. Epub 2019 Feb 11. PMID 30968152
- [Result] Sandur SK, Deorukhkar A, Pandey MK, Pabon AM, Shentu S, Guha S, Aggarwal BB, Krishnan S. Curcumin modulates the radiosensitivity of colorectal cancer cells by suppressing constitutive and inducible NF-kappaB activity. Int J Radiat Oncol Biol Phys. 2009 Oct 1;75(2):534-42. doi: 10.1016/j.ijrobp.2009.06.034. PMID 19735878
- [Result] Arun P, Sagayaraj A, Azeem Mohiyuddin SM, Santosh D. Role of turmeric extract in minimising mucositis in patients receiving radiotherapy for head and neck squamous cell cancer: a randomised, placebo-controlled trial. J Laryngol Otol. 2020 Feb 7:1-6. doi: 10.1017/S0022215120000316. Online ahead of print. PMID 32029014
- [Result] Antony B, Merina B, Iyer VS, Judy N, Lennertz K, Joyal S. A Pilot Cross-Over Study to Evaluate Human Oral Bioavailability of BCM-95CG (Biocurcumax), A Novel Bioenhanced Preparation of Curcumin. Indian J Pharm Sci. 2008 Jul-Aug;70(4):445-9. doi: 10.4103/0250-474X.44591. PMID 20046768
- [Result] Shehzad A, Wahid F, Lee YS. Curcumin in cancer chemoprevention: molecular targets, pharmacokinetics, bioavailability, and clinical trials. Arch Pharm (Weinheim). 2010 Sep;343(9):489-99. doi: 10.1002/ardp.200900319. PMID 20726007
- [Result] Ismail NI, Othman I, Abas F, H Lajis N, Naidu R. Mechanism of Apoptosis Induced by Curcumin in Colorectal Cancer. Int J Mol Sci. 2019 May 17;20(10):2454. doi: 10.3390/ijms20102454. PMID 31108984
- [Result] Jurenka JS. Anti-inflammatory properties of curcumin, a major constituent of Curcuma longa: a review of preclinical and clinical research. Altern Med Rev. 2009 Jun;14(2):141-53. PMID 19594223

DOCUMENTS (1):
  • Study Protocol (2025-11-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT07248020/Prot_000.pdf